CLINICAL TRIAL: NCT04840602
Title: A Phase II Randomized Study Comparing Ibrutinib and Rituximab vs. Venetoclax and Rituximab in Previously Untreated Waldenström's Macroglobulinemia (WM) / Lymphoplasmacytic Lymphoma (LPL)
Brief Title: Testing the Combination of Venetoclax and Rituximab, in Comparison to the Usual Treatment (Ibrutinib and Rituximab) for Waldenstrom's Macroglobulinemia/Lymphoplasmacytic Lymphoma
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Other - For RRA for Venetoclax issued 10/17/2025
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-02851; NCI-2021-02851 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S2005 (Other: SWOG); S2005 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2021-04-09; First posted 2021-04-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-11

CONDITIONS: Lymphoplasmacytic Lymphoma; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Waldenstrom Macroglobulinemia | interventions — Specimen Handling; Biopsy; ibrutinib; Magnetic Resonance Spectroscopy; Rituximab; CT-P10; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (ibrutinib, rituximab) (Active Comparator): Patients receive ibrutinib PO QD on days 1-28 of cycles 1-24 and rituximab IV on days 1, 8, 15, and 22 of cycles 2 and 5. Cycles repeat every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients with progressive disease during Arm I may receive rituximab and venetoclax as in Arm II for up to an additional 24 cycles. Patients undergo CT or PET/CT and bone marrow biopsy and aspiration as well as blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Ibrutinib; Procedure: Positron Emission Tomography; Biological: Rituximab
- Arm II (venetoclax, rituximab) (Experimental): Patients receive venetoclax PO QD on days 1-28 of each cycle and rituximab IV on days 1, 8, 15, and 22 of cycles 2 and 5. Cycles repeat every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients with progressive disease during Arm II may receive ibrutinib and rituximab as in Arm I for up to an additional 24 cycles. Patients undergo CT or PET/CT and bone marrow biopsy and aspiration as well as blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Biological: Rituximab; Drug: Venetoclax

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow biopsy and aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and aspiration
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA 032765; CRA-032765; CRA032765; Imbruvica; PCI 32765; PCI-32765; PCI32765
  Arms: Arm I (ibrutinib, rituximab)
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Biological: Rituximab — Given IV
  Other Names: ABP 798; ABP-798; ABP798; BI 695500; BI-695500; BI695500; Blitzima; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT P10; CT-P10; CTP10; GP 2013; GP-2013; GP2013; IDEC 102; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; IDEC102; Ikgdar; Mabtas; MabThera; Monoclonal Antibody IDEC-C2B8; PF 05280586; PF-05280586; PF05280586; Riabni; Ritemvia; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar GP2013; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-blit; Rituximab-pvvr; Rituximab-rite; Rituximab-rixa; Rituximab-rixi; Rixathon; Riximyo; RTXM 83; RTXM-83; RTXM83; Ruxience; Truxima
Drug: Venetoclax — Given PO
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto
  Arms: Arm II (venetoclax, rituximab)

SUMMARY:
This phase II trial studies the effects of venetoclax and rituximab in comparison to ibrutinib and rituximab in treating patients with previously untreated Waldenstrom's macroglobulinemia/lymphoplasmacytic lymphoma. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Rituximab is a monoclonal antibody. It binds to a protein called CD20, which is found on B cells (a type of white blood cell) and some types of cancer cells. This may help the immune system kill cancer cells. Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Giving venetoclax and rituximab may work better in treating patients with previously untreated Waldenstrom's macroglobulinemia than ibrutinib and rituximab alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the rate of very good partial response or better (VGPR or better) in previously untreated participants with Waldenström's macroglobulinemia (WM)/lymphoplasmacytic lymphoma (LPL) who are treated upfront with ibrutinib plus rituximab (IR) versus (vs.) venetoclax plus rituximab (VR) regimen.

SECONDARY OBJECTIVES:

I. To compare overall response rates (ORR) in WM participants treated upfront with IR vs. those treated with VR.

II. To compare progression-free survival (PFS), time to next treatment, duration of response in WM participants treated upfront with IR vs. those treated with VR.

III. To compare the rate of complete response (CR) in WM participants treated upfront with IR vs. those treated with VR.

IV. To evaluate the safety of the IR regimen as compared to VR regimen in participants with WM.

V. To evaluate the time to VGPR in WM participants treated upfront with IR and those treated with VR.

VI. To evaluate the ORR in participants who progress on treatment with IR and VR and are crossed over to the other respective arm.

VII. To compare overall survival (OS) in WM participants treated upfront with IR vs. those treated with VR.

BANKING OBJECTIVE:

I. To bank specimens for future correlative studies.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive ibrutinib orally (PO) once daily (QD) on days 1-28 of cycles 1-24 and rituximab intravenously (IV) on days 1, 8, 15, and 22 of cycles 2 and 5. Cycles repeat every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients with progressive disease during Arm I may receive rituximab and venetoclax as in Arm II for up to an additional 24 cycles. Patients undergo computed tomography (CT) or positron emission tomography (PET)/CT and bone marrow biopsy and aspiration as well as blood sample collection throughout the trial.

ARM II: Patients receive venetoclax PO QD on days 1-28 of each cycle and rituximab IV on days 1, 8, 15, and 22 of cycles 2 and 5. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients with progressive disease during Arm II may receive ibrutinib and rituximab as in Arm I for up to an additional 24 cycles. Patients undergo CT or PET/CT and bone marrow biopsy and aspiration as well as blood sample collection throughout the trial.

After completion of study treatment, patients removed from protocol prior to progression are followed every 3 months until progression, death or 5 years after initial registration, whichever occurs first. Patients followed after progression of disease are followed every 6 months until death or 5 years after initial registration.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have had a confirmed diagnosis of Waldenstrom's macroglobulinemia (WM)/lymphoplasmacytic lymphoma (LPL). Participants must have measurable disease as determined by IgM protein quantification.

  * IgM Spike: ≥ 500 mg/dL (≥ 5 g/L)
  * Extramedullary disease: The manifestation of a lymphoid mass outside of the bone marrow, resulting in enlargement in extramedullary organs such as the lymph nodes or spleen. Note: all participants must have measurable IgM spike, but are not required to have extramedullary disease
* Testing to establish baseline disease status must be performed within 28 days prior to registration
* Participants must have at least one of the criteria to require therapy for WM including anemia, thrombocytopenia, neuropathy related to WM, symptomatic hyperviscosity or serum viscosity levels greater than 4.0 centipoises, WM associated glomerulonephritis or renal disease, bulky disease, or constitutional symptoms. Constitutional symptoms can be described as unintentional weight loss >= 10% within the previous 6 months prior to screening; Fevers higher than 100.5 degrees Fahrenheit (F) or 38.0 degrees Celsius (C) for 2 or more weeks prior to screening without evidence of infection; Night sweats for more than 1 month prior to screening without evidence of infection; Clinically relevant fatigue which is not relieved by rest due to WM
* Participants who require ongoing use or received a moderate or strong CYP3A inducer, moderate or strong CYP3A inhibitor, P-gp inhibitor within 7 days prior to the first dose of study drug will be excluded from the study. If such participants can be safely switched to an alternative agent, then the participants will be eligible to enroll
* Participants must not have had prior systemic therapy. Prior therapy with rituximab will be allowed as long as the last rituximab dose was at least 6 months prior to registration
* Participants must be >= 18 years of age
* Participants must have history and physical exam within 28 days prior to registration
* Participants must have Zubrod performance status =< 2
* Participants must have evidence of adequate renal function, as defined by creatinine clearance (CrCl) >= 30 mL/min. Values must be obtained within 14 days prior to registration
* Total bilirubin =< 1.5 x IULN (institutional upper limit of the norm) (within 14 days prior to registration)
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) =< 3 x IULN (within 14 days prior to registration)
* Alkaline phosphatase =< 3 x IULN (within 14 days prior to registration)
* Platelet count >= 50,000 cells/mm^3 (within 14 days prior to registration)

  * NOTE: Transfusion and/or growth factor support is allowed up to 7 days prior to registration
* Hemoglobin >= 7.5 g/dL (within 14 days prior to registration)

  * NOTE: Transfusion and/or growth factor support is allowed up to 7 days prior to registration
* Absolute neutrophil count (ANC) >= 1,000 cells/mm^3 (within 14 days prior to registration)

  * NOTE: Transfusion and/or growth factor support is allowed up to 7 days prior to registration
* Participants with known human immunodeficiency virus (HIV)-infection are eligible providing they are on effective anti-retroviral therapy and have undetectable viral load at their most recent viral load test and within 6 months prior to registration
* Participants must be able to take and swallow oral medication (capsules) whole. Participants may not have any known impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of the study drug (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* Participants must not be intolerant to rituximab
* Participants must not have known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding localized skin and nail bed fungal infections) at study enrollment, or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) 4 weeks prior to registration
* Participants must not be seropositive for hepatitis C (except in the setting of sustained virologic response, defined as undetectable viral load at least 12 weeks after completion of antiviral therapy). Hepatitis C virus (HCV) testing is only required if clinically indicated or if the participant has a history of HCV
* Participants must not consume grapefruit, Seville oranges or starfruit within 3 days prior to the first dose of venetoclax
* Participants must not be pregnant or nursing because venetoclax has not been studied in pregnant or nursing women and the mechanism of action is expected to cause fetal harm. A woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months. In addition to routine contraceptive methods, "effective contraception" e.g., implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], complete abstinence, or sterilized partner) and a barrier method (e.g., condom, cervical ring, sponge, etc.). This also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation. However, if at any point a previously celibate participant chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures throughout the study and for at least 30 days after competition of therapy
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the participant is currently in complete remission, or any other cancer from which the participant has been disease free for two years or watchful waiting is appropriate in the opinion of the treating physician. Also, malignancy that in the opinion of the investigator, is considered cured with minimal risk of recurrence within 5 years, is permissible consideration of eligibility for this trial
* Participants must be offered the opportunity to participate in specimen banking
* Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines. For participants with impaired decision-making capabilities, legally authorized representatives may sign and give informed consent on behalf of study participants in accordance with applicable federal, local, and Central Institutional Review Board (CIRB) regulations
* As a part of the Oncology Participant Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* CROSSOVER CRITERIA: Participants must have been registered and received treatment in the IR or VR arm and must show progression of disease at any time during cycles 3-24
* CROSSOVER CRITERIA: In case of transformation to intermediate or high-grade lymphoma or development of Bing-Neel syndrome the participants will not undergo registration step 2 crossover and will be taken off the study
* CROSSOVER CRITERIA: Participants must have Zubrod performance status =< 2
* CROSSOVER CRITERIA: Participants must have evidence of adequate renal function, as defined by creatinine clearance (CrCl) >= 30 mL/min. Values must be obtained within 14 days prior to registration
* CROSSOVER CRITERIA: Participants must have no evidence of marked hepatic dysfunction on any recent liver function tests within 14 days prior to registration
* CROSSOVER CRITERIA: Platelet count >= 50,000 cells/mm^3 (without within 14 days prior to registration)

  * NOTE: Transfusion and/or growth factor support is allowed up to 7 days prior to registration
* CROSSOVER CRITERIA: Hemoglobin >= 7.5 g/dL (without within 14 days prior to registration)

  * NOTE: Transfusion and/or growth factor support is allowed up to 7 days prior to registration
* CROSSOVER CRITERIA: Absolute neutrophil count (ANC) >= 1,000 cells/mm^3 (without within 14 days prior to registration)

  * NOTE: Transfusion and/or growth factor support is allowed up to 7 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Very good partial response or better (VGPR or better) rate | Up to 5 years
  A Cochran-Mantel-Haenszel test will be performed to compare the VGPR or better rates in Arm 1 and Arm 2 accounting for the stratification factor of prior rituximab, and VGPR or better rate will be reported in each study arm with a binomial confidence interval.

SECONDARY OUTCOMES:
Progression-free survival | From the date of registration to the date of first documentation of progressive disease or symptomatic deterioration, or death due to any cause, assessed up to 5 years
  Will be analyzed using the Kaplan-Meier method, and a stratified log-rank test will be performed to compare survival outcomes in the ibrutinib rituximab (IR) and venetoclax rituximab (VR) arms while controlling for the effects from the stratification factor of prior rituximab treatment.
Overall survival | From the date of registration to the date of death due to any cause, assessed up to 5 years
  Will be analyzed using the Kaplan-Meier method, and a stratified log-rank test will be performed to compare survival outcomes in the IR and VR arms while controlling for the effects from the stratification factor of prior rituximab treatment.
Rate of complete response | From the date of registration to the date of complete response, assessed up to 5 years
  Will be analyzed using the cumulative incidence competing risks method.
Overall response rate | Up to 5 years
  Defined as the percentage of participants achieving a best response of complete response, very good partial response, or partial response while on study. Will be reported with a binomial confidence interval.
Time to VGPR or better | Up to 5 years
  Defined as the percentage of participants achieving a best response of very good partial response or better while on study. Will be reported with a binomial confidence interval.
Incidence of adverse events | Up to 5 years
  As assessed by Common Terminology Criteria for Adverse Events Version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Sikander Ailawadhi, Principal Investigator — SWOG Cancer Research Network
Locations (113):
- United States (113):
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Centralia Oncology Clinic, Centralia, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Levine Cancer Institute-Gaston, Gastonia, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Central Ohio Breast and Endocrine Surgery, Gahanna, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm